CLINICAL TRIAL: NCT06975020
Title: CANBiome: Pilot-Study for the Comparison of Biomarkers Between Regular Cannabis Users and Non-Users
Brief Title: Pilot-Study for the Comparison of Biomarkers Between Regular Cannabis Users and Non-Users
Acronym: CANBiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University Psychiatric Clinics Basel, University of Basel, Basel, Switzerland (Unknown); Department of Endocrinology, Diabetology and Metabolism, University Hospital Basel, Basel, Switzerland (Unknown); Biopharmacy, Department of Pharmaceutical Sciences, University of Basel, Basel, Switzerland (Unknown); Institute of Forensic Medicine, University of Basel, Basel, Switzerland (Unknown)
Responsible Party: Principal Investigator, Urs Duthaler, PD Dr., University of Basel
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-00354
Record Dates: First submitted 2025-04-11; First posted 2025-05-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Driving Under the Influence of Cannabis
Keywords: Cannabis; Driving; Biomarker
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis group (Experimental)
  Interventions: Drug: Participants will prepare their cannabis product ad libitum and inhale the prepared product as usual for a maximum of 15 minutes.
- Control group (No Intervention)

INTERVENTIONS:
Drug: Participants will prepare their cannabis product ad libitum and inhale the prepared product as usual for a maximum of 15 minutes. — Participants will prepare and inhale their cannabis product ad libitum for a maximum of 15 minutes. Prior to inhaling cannabis (the baseline), and for three hours thereafter, biological samples (e.g., blood) will be collected. Participants will be asked to complete a series of questionnaires addressing their (subjective) neurocognitive function and well-being, as well as their self-rated driving ability and subjective cannabis effects.
  Arms: Cannabis group

SUMMARY:
The relevance of driving under the influence of cannabis is becoming increasingly important in the context of legalization. However, the measurement of tetrahydrocannabinol (THC) blood concentration is an inadequate marker for assessing driving impairment. Currently, there is no reliable marker available for estimating the time of last cannabis inhalation, which would provide a promising tool for regulating driving under the influence of cannabis. This pilot study aims to explore potential biomarkers and factors that could approximate the timing of the last cannabis inhalation, with emphasis on the potential explanation of interindividual differences in THC pharmacokinetics and -dynamics. The results will assist future research aimed at improving the ability to distinguish between impaired and unimpaired cannabis users in road traffic. These findings are of significant importance for road safety and for society at large, as they may provide more objective markers for cannabis inhalation, thereby permitting a methodologically sound evaluation of driving under the influence of cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Experience of smoking cannabis products, on average once a week. This may be in combination with tobacco.
* Age 18-65 years Possession of driving license in at least one of the categories A, B, A1; B1, F, G or M
* Sufficient knowledge of German
* No cannabis inhalation or nicotine consumption on study day
* No alcohol consumption within the last 24 h

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Current or previous major psychiatric disorder (e.g., major depression, schizophrenia spectrum disorder)
* Pregnancy or breastfeeding
* Intake of CYP2C9, CYP2C19, and CYP3A4-inducers in the last 4 weeks before the study visit, e.g. rifampicin (antibiotic), carbamazepine (anticonvulsant), phenobarbital (anticonvulsant), phenytoin (anticonvulsant) or inhibitors, such as amiodarone (class III antiarrhythmic medication), antifungal drugs such as fluconazole, miconazole, voriconazole and itraconazole, antibiotics such as clarithromycin and sulfamethoxazole, ritonavir (protease inhibitor) and grapefruit juice.
* The following conditions: vasopressin deficiency, pituitary tumor, active malignancy, severe hyponatremia requiring treatment, congestive heart failure, liver cirrhosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of phytochemicals in cannabis sativa (e.g. cannabinoids and flavonoids) and their metabolites in human whole blood samples. | 24 months
  Quantification of the blood concentration of cannabis sativa phytochemicals such as minor cannabinoids, cannabinoids, and flavonoids. Blood samples will be analyzed at baseline and several time-points (0, 10, 20, 60, 180) post consumption of cannabis. Concentrations will be reported as ng/mL whole blood.

SECONDARY OUTCOMES:
Measurement of the expression levels of relevant genes e.g. cannabinoid receptor 1 (CB1) and cannabinoid receptor 2 (CB2) in whole blood samples by e.g. RT-PCR to evaluate especially their correlation with cannabinoid plasma levels, metabolism, and ph | 24 months
Assessment of selected genetic polymorphisms in the genes known to interact with cannabinoids (i.e. CYP2C9, CYP2C19) by e.g. RT-PCR to evaluate their influence on cannabinoid plasma levels and the ability to predict cannabinoid metabolism and pharmaco | 24 months
Quantitation of biomarkers applicable to determine the activity of enzymes or transporters known to be involved in the handling of cannabinoids (e.g. 4-ß-hydroxycholesterol, Coproporphyrin I und Coproporphyrin III) | 24 months
Comparison of DNA methylation profiles on blood-derived DNA samples between regular and non-cannabis users by evaluating key CpG sites (e.g., in the MCU gene) that interplay with risk factors and mental health by e.g. targeted Illumina DNA methylation | 24 months
Analysis of the protein-bound and free fractions of the different cannabinoids and their metabolites using e.g. equilibrium dialysis or ultracentrifugation | 24 months
Targeted and untargeted analysis of endogenous biomarkers (e.g. endocannabinoids) using e.g. high-resolution mass-spectrometry | 24 months
Subjectively experienced effects of cannabis inhalation (e.g. subjective driving ability, psychological effects and well-being) assessed by questionnaires (e.g. VAS) | 24 months
The effects of cannabis inhalation on neurocognition by non-invasive, neurocognitive testing | 24 months
Self-reported mood as measured e.g. by the Bf-SR questionnaire. | 24 months
Usual reasons for cannabis use as measured e.g. by the Marijuana Motives Questionnaire (MMQ) | 24 months
Measurement of hormones and biomarkers involved in the regulation of fluid balance (e.g. plasma osmolality …) | 24 months
Measurement of hormones and biomarkers of the anterior and posterior pituitary gland (e.g., plasma oxytocin, neurophysin I, ACTH, TSH, prolactin …) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of forensic medicine, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kraemer M, Madea B, Hess C. Detectability of various cannabinoids in plasma samples of cannabis users: Indicators of recent cannabis use? Drug Test Anal. 2019 Oct;11(10):1498-1506. doi: 10.1002/dta.2682. Epub 2019 Sep 1. PMID 31407526
- [Background] Berman P, Futoran K, Lewitus GM, Mukha D, Benami M, Shlomi T, Meiri D. A new ESI-LC/MS approach for comprehensive metabolic profiling of phytocannabinoids in Cannabis. Sci Rep. 2018 Sep 24;8(1):14280. doi: 10.1038/s41598-018-32651-4. PMID 30250104
- [Background] Manthey J, Freeman TP, Kilian C, Lopez-Pelayo H, Rehm J. Public health monitoring of cannabis use in Europe: prevalence of use, cannabis potency, and treatment rates. Lancet Reg Health Eur. 2021 Sep 24;10:100227. doi: 10.1016/j.lanepe.2021.100227. eCollection 2021 Nov. PMID 34806072
- [Background] Marcotte TD, Umlauf A, Grelotti DJ, Sones EG, Sobolesky PM, Smith BE, Hoffman MA, Hubbard JA, Severson J, Huestis MA, Grant I, Fitzgerald RL. Driving Performance and Cannabis Users' Perception of Safety: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Mar 1;79(3):201-209. doi: 10.1001/jamapsychiatry.2021.4037. PMID 35080588